CLINICAL TRIAL: NCT01638156
Title: Arterial Stiffness and Wave Reflections as Determinants of Regression of Left Ventricular Hypertrophy and Fibrosis Assessed With Cardiac MRI After Aortic Valve Replacement for Severe Aortic Stenosis
Brief Title: Cardiac MRI for Severe Aortic Stenosis
Status: Completed | Type: Observational
Sponsor: American College of Radiology (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: ACRIN PA 4008
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Aortic Stenosis
Keywords: Aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collecting three tubes of blood: 10-mL of blood for plasma sampling, 10-mL of serum, and a microtube or other adequate sample for hematocrit measurements. Hematocrit measurements within 24 hours prior to the cardiac MRI scan. Serum and plasma samples will be stored at -80°C in 0.5 mL vials.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will evaluate the importance of arterial stiffness and wave reflections as determinants of persistent left ventricular (LV) hypertrophy and fibrosis (assessed using cardiac magnetic resonance imaging [MRI]) after correction of severe stenosis of the aortic valve. The hypothesis will test whether stiff arteries and increased wave reflections impede pumping of blood by the LV after aortic valve replacement (AVR)and precent adequate regression (improvement) of hypertrophy and fibrosis of the myocardium despite correction of aortic valve stenosis.

DETAILED DESCRIPTION:
A total of 80 participants will be enrolled into the study from site with the protocol-required technology. The Pennsylvania Department of Health funding for this trial is limited to sites in Pennsylvania. Participants will undergo pre- and post-operative cardiac MRI, blood draws, a 6-minute walk test, arterial tonometry, medical history assessment, and quality-of-life questionnaires to characterize the pathophysiologic factors causing variability in regression after AVR. Researchers will evaluate the role of specific hemodynamic abnormalities as determinants of post-AVR LV remodeling (LV hypertrophy and LV myocardial fibrosis) as seen on contrast-enhanced cardiac MRI. The trial also will evaluate a non-contrast-enhanced MRI approach (T1rho) potentially effective in assessing LV myocardial fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Severe symptomatic aortic stenosis (estimated aortic valve area <1 cm2) 1,2 as documented on a transthoracic echocardiogram (ECG) performed within 4 months prior to enrollment
* Planned for AVR within 8 weeks after enrollment
* Able to have a cardiac MRI within 3 weeks prior to the AVR surgery
* A preoperative coronary angiography demonstrating the absence of hemodynamically-significant CAD in need of revascularization during AVR surgery
* Able to tolerate cardiac MRI with gadolinium contrast as required by protocol, to be performed at an ACRIN-qualified facility using an ACRIN-qualified MR scanner
* Willing and able to provide a written informed consent

Exclusion Criteria:

* Not suitable to undergo cardiac MRI or use the contrast agent gadolinium because of:

  * Claustrophobia
  * Presence of metallic objects or implanted medical devices in body (i.e., implanted cardiac pacemaker or defibrillator, central nervous system aneurysm clips, implanted neural stimulators, cochlear implant, ocular foreign body [e.g., metal shavings], other implanted medical devices [e.g., drug infusion port], insulin pump, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants)
  * Weight greater than that allowable by the MRI table
* Known LV ejection fraction <50%
* Previous aortic valve surgery
* Planned additional valve repair/replacement
* Infective endocarditis
* Moderate or severe aortic valve regurgitation
* Rhythm other than sinus rhythm (i.e., atrial fibrillation) that results in an irregular heartbeat, compromising the quality of MRI and tonometry data acquisition, as documented on an ECG performed within 8 weeks prior to enrollment
* Presence of hemodynamically-significant CAD that would require revascularization during the AVR surgery
* Myocardial infarction or unstable angina in the previous month
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 of body surface area documented within 4 weeks prior to enrollment

NOTE: This threshold has been deemed appropriate for this study, rather than <30 mL/min/1.73m2, since eGFR is likely to decrease for participants between the baseline and 6-month examinations. The protocol calls for gadolinium administration in the 6-month evaluation, and gadolinium administration is contraindicated in the presence of an eGFR <30 mL/min/1.73m2. Therefore, initially excluding patients who have an eGFR < 60 mL/min/1.73m2 will minimize the presence of an eGFR <30 mL/min/1.73m2 at the time of the 6-month evaluation.

An eGFR < 30 mL/min/1.73m2 of body surface area or acute kidney injury will be a contraindication to gadolinium contrast administration, and participants with insufficient kidney function immediately before the 6-month cardiac MRI will undergo an MRI without contrast-enhancement and will continue on-study.

* Presence of a bicuspid aortic valve, which is associated with an intrinsic aortopathy that may affect arterial load in its own right;
* Resting heart rate >120 beats per minute, systolic blood pressure >180 mm Hg, or diastolic blood pressure > 100 mm Hg
* Pregnancy or intent to become pregnant
* Conditions that would make the study measurements less accurate or unreliable (i.e., frequent premature beats that may affecting cardiac gating, anatomic neck characteristics impeding arterial tonometry, inability to perform an adequate breath hold for cardiac MRI acquisitions) or the reliable post-operative follow-up of patients (for at least 6 months post-AVR) unlikely
* Known peripheral vascular disease, which may limit the ability to exercise independently of cardiac status due to claudication
* Unwillingness of the patient to undergo a cardiac MRI
* Unwillingness of the patient to sign the consent form
* Any condition limiting life expectancy to <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 years of age or older with no contraindications to gadolinium contrast-enhanced MRI of the heart who are able to have a cardiac MRI in the 21 days before the AVR operation, have been diagnosed with severe symptomatic aortic stenosis (estimated aortic valve area <1 cm2),1,2 and are scheduled for AVR between 0 and 28 days after enrollment. Potential participants will have undergone a clinically indicated pre-operative evaluation showing the absence of hemodynamically-significant CAD that would require revascularization during the AVR operation.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiac MRI before and after to detect changes in response to aortic valve replacement (AVR) for sever aortic stenosis. | 1-2 years
  To test the hypothesis that increased stiffness of the aortic wall and arterial wave reflections correlate with an adequate regression (improvement) of LV hypertrophy and LV myocardial fibrosis measured with cardiac MRI after AVR for severe aortic stenosis.

SECONDARY OUTCOMES:
Evaluate role of specific hemodynamic abnormalities that depend on systemic arteries, as determinants of post-AVR improvement in left ventricular (LV) remodeling (LV hypertrophy and LV myocardial fibrosis) | 1-2 years
  To test the hypothesis that increased stiffness of the aortic wall and increased arterial wave reflections are important determinants of LV hypertrophy and LV myocardial fibrosis in participants with severe aortic stenosis.
Myocardial T1rho mapping | 1-2 years
  To test the hypothesis that myocardial T1rho mapping, a novel myocardial tissue characterization MRI technique, correlates with LV myocardial fibrosis assessed with post-gadolinium myocardial T1 measurements in participants with severe aortic stenosis.
Changes in myocardial T1rho after AVR | 1-2 years
  To test the hypothesis that changes in myocardial T1rho after AVR in participants with severe aortic stenosis correlates with changes in LV myocardial fibrosis assessed with post-gadolinium myocardial T1 measurements.
Stiffness and reflection correlates with physical fitness after AVR | 1-2 years
  To test the hypothesis that increased stiffness of the aortic wall and arterial wave reflections correlate with physical fitness (assessed via a 6-minute walk test) after AVR for severe aortic stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Akers, MD, PhD, Study Chair — Philadelphia Veterans Administration Medical Center; Julio A. Chirinos, MD, Study Chair — Philadelphia Veterans Administration Medical Center
Locations (2):
- United States (2):
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania